## The Role of Matrix Metalloproteinase 2 and 9 Enzymes in Developing Chronic Thromboembolic Pulmonary Hypertension

(NCT04773028)

Date: 3 March 2020

## **Statistical Analysis**

In this prospectively planned study, the data of 24 patients who were operated for CTEPH and 24 patients who underwent lobectomy or pneumonectomy, a total of 48 patients will be evaluated. Power analysis was used to determine the number of patients, the number of people was calculated as 48 people, 24 cases and 24 controls, with 97% effect size, 95% confidence and 5% acceptable error. The data were analyzed with the SPSS package program. Continuous variables are given as mean ± standard deviation, categorical variables as numbers and percentages. When parametric test assumptions are provided in independent group comparisons, the Significance Test of the Difference Between Two Means; If parametric test assumptions were not provided, Mann Whitney U and Kruskal Wallis tests were used, and Chi-square analysis was used for comparison of categorical variables. The relationship between variables was analyzed using Spearman for nonparametric variables and Pearson correlation analysis for parametric variables. p ≤ 0.05 was considered significant.